CLINICAL TRIAL: NCT03403387
Title: Effects of Shield Nutraceuticals GlutenShield on Short Chain Fatty Acid Production, Gut Microbiota, and Markers of Inflammation in Individuals With GI Symptoms
Brief Title: Effects of GlutenShield, a Prebiotic, Probiotic, and Enzyme Supplement, on the Gut Microbiome of Adults With GI Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Tennessee State University (Other)
Collaborators: East Tennessee State University, College of Clinical and Rehabilitative Health Sciences (Unknown); East Tennessee State University, College of Public Health, Department of Health Sciences (Unknown); Shield Nutraceuticals (Unknown)
Responsible Party: Principal Investigator, Kaitlyn Webb, Graduate Student in Clinical Nutrition, East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1117.22f
Record Dates: First submitted 2018-01-05; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Gastrointestinal Symptoms

STUDY DESIGN:
Intervention Model Description: Half of the participants will be randomized to receive the supplement and the other half will receive the placebo.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlutenShield (Experimental): 3 capsules of GlutenShield supplement/day for 28 days
  Interventions: Dietary Supplement: GlutenShield
- Placebo (Placebo Comparator): 3 capsules of the placebo (Avicel and bentonite powder (for color))/ day for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GlutenShield — combination probiotic, prebiotic, and enzyme supplement
  Arms: GlutenShield
Other: Placebo — Avicel (cellulose) and bentonite powder
  Arms: Placebo

SUMMARY:
This study evaluates the effects of combination probiotic, prebiotic, and enzyme supplementation on the colonic microbiome of individuals with GI symptoms (e.g. diarrhea, constipation, increased gas). Half of the participants will receive the placebo while the other half will receive the supplement for 28 days.

DETAILED DESCRIPTION:
The purpose of this research is to identify if there is a relationship between GlutenShield, a combination prebiotic, probiotic, and enzyme supplement, and the gut environment.

The study will be a split, 28-day randomized, partially blinded design. Subjects will be randomly assigned to one of two groups. One group will complete a 28-day treatment period with GlutenShield taken 3x/day with meals. The other group will complete a 28-day placebo period with the placebo taken 3x/day with meals. The placebo will contain Avicel (cellulose) and bentonite powder (to have a similar color as GlutenShield). Participants will be blinded to which group/ treatment they are being given. Serum and fecal samples will be collected at baseline and on day 29. Participants will also complete a gastrointestinal symptoms questionnaire, a food frequency questionnaire and a psychosocial measures of self questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who express gastrointestinal symptoms more than three times per week as identified through the Gastrointestinal Symptom Questionnaire (such as abdominal pain/ discomfort, heartburn, acid regurgitation, bloating, nausea and vomiting, abdominal distention, eructation (burping), increased gas, decreased passage of stools, increased passage of stools, loose stools, hard stools, urgent need for defecation, or feeling of incomplete evacuation)
* Healthy with few health complications
* Adults ages 18 or older

Exclusion Criteria:

* Anyone under the age of 18
* Individuals diagnosed with celiacs, IBS, Crohn's disease, ulcerative colitis, or short bowel syndrome
* Individuals who have previously taken GlutenShield
* Individuals who are currently taking prebiotics, probiotics, enzymes, non-steroidal anti-inflammatory drugs, fish oil, and/or fiber supplements (unless use is halted in the voluntary 2-week washout period prior to the study)
* Individuals who are pregnant or intend to become pregnant during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-22 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fermentation Profile- Short Chain Fatty Acid Concentration | Baseline and Day 29
  Measuring change short chain fatty acid concentrations in fecal matter (analyzed using gas chromatography) from baseline to after 28 days.
Change in Microbial Population and Concentration | Baseline and Day 29
  Measuring change from baseline of fecal microbial populations and concentrations (using genomic sequencing).
Change in Inflammation | Baseline and Day 29
  Measuring change in serum markers of inflammation (IgA and IgG, GM-CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, TNF-α) over 28 days. Values will be used to determine a change in overall inflammatory status.

SECONDARY OUTCOMES:
Dietary Intake | Baseline
  Identifying typical dietary intake over the past month using Block Food Frequency Questionnaire
Physical Activity | Baseline
  Identifying typical physical activity over the past month using Block Food Frequency Questionnaire
Change in Oxidative Stress | Baseline and Day 29
  Measuring changes in serum markers of oxidative stress (8-isoprostaglandin F2a)
Changes in Psychosocial Measures of Self | Baseline and Day 29
  Measuring changes in psychosocial measures of self (Profile of Mood States 2nd Edition survey)
Changes in Adipokine Response | Baseline and Day 29
  Measuring changes in adipokine response (Bio-Plex Pro Human Diabetes Adipsin and Adiponectin assays)

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn Webb, BS, Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data. Data will be de-identified.